CLINICAL TRIAL: NCT04178174
Title: Stereotactic Boost and SHOrt-course Radiation Therapy for HPV-associated OroPharynx Cancer Trial: A Randomized Multicentric Phase III Trial
Brief Title: Stereotactic Boost and Short-course Radiation Therapy for Oropharynx Cancer
Acronym: SHORT-OPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: M.D. Anderson Cancer Center (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Houda Bahig, Radiation Oncologist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHORT-OPC
Record Dates: First submitted 2019-11-17; First posted 2019-11-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Oropharynx Cancer; Human Papilloma Virus
Keywords: head and neck cander; Oropharynx cancer; Human papilloma virus; Radiotherapy; Stereotactic body radiotherapy; Chemotherapy; De-intensification
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SABR boost and de-escalated chemoradiation (Experimental): SABR boost of 14 Gy in 2 fractions to the GTV, immediately followed by de-escalated chemoradiation. De-escalated chemoradiation will consist in 40 Gy in 20 fractions with concurrent high dose Cisplatin (3-weekly, 100 mg/m2) for 2 cycles, aiming for a cumulative dose of 200 mg/m2.
  Interventions: Radiation: SABR boost and de-escalated chemoradiation
- Standard chemoradiation (Active Comparator): The standard arm will consist of conventionally radiation to a dose of 70 Gy in 33 fractions concurrently with high dose Cisplatin (3-weekly, 100 mg/m2) for 2-3 cycles, aiming for a cumulative dose of ≥ 200 mg/m2.
  Interventions: Radiation: Standard chemoradiation

INTERVENTIONS:
Radiation: SABR boost and de-escalated chemoradiation — Stereotactic body radiotherapy boost to the gross tumor volume to a dose of 14 Gy in 2 fractions, followed by cisplatin-based chemoradiation to a dose of 40 Gy in 20 fractions
  Arms: SABR boost and de-escalated chemoradiation
Radiation: Standard chemoradiation — Standard Cisplatin-based chemoradiation to a dose of 70 Gy in 33 fractions
  Arms: Standard chemoradiation

SUMMARY:
This is a randomized clinical trial comparing the outcomes of short-course chemoradiation consisting in stereotactic boost to the gross tumor and de-esclalated chemoradiation to the elective neck in human papilloma associated oropharynx cancer vs. the current standard 7-week course chemoradiation.

DETAILED DESCRIPTION:
Concurrent platinum-based chemoradiation remains the standard of care in locally advanced head and neck cancer. The current standard radiation regimen consists in a 7-week course of conventionally fractionated radiotherapy to the gross tumor volume (GTV), along with bilateral prophylactic neck irradiation to an elective dose of ~ 50 Gy in 2 Gy per fraction. In addition to being cumbersome, the current protracted daily radiation course is associated with high rates of acute and late toxicities and significant deterioration of patients' quality of life. In the light of the remarkably improved prognosis of the distinct subgroup of HPV-OPC, there is growing interest for treatment de-intensification strategies in contemporaneous OPC cohorts.

Stereotactic ablative radiotherapy (SABR) allows for ultra-precise delivery of ablative radiation dose over a small number of fractions, by combining sharp dose gradients with use of optimal image guidance. The increased conformity and reduced margins used in SABR can substantially reduce the dose to surrounding organs at risk and could therefore reduce toxicity. In addition, previous work has shown that an elective dose of 40 Gy in 2 Gy per fraction, in conjunction with chemotherapy, is sufficient for microscopic sterilisation of cancer cells and can translate into a reduction of toxicities.

The goal of this trial is to compare the efficacy and safety of short-course chemoradiation consisting in stereotactic boost to the gross tumor of 14 Gy in 2 fractions followed by de-esclalated chemoradiation (40 Gy in 20 fractions and concurrent 2 cycles of Cisplatin 100mg/m2) in human papilloma associated oropharynx cancer vs. the current standard 7-week course chemoradiation (70 Gy in 33 fractions with 2-3 cycles of Cisplatin 100mg/m2).

This is an open label randomized phase III non inferiority trial. Patients will be randomized using a 1:1 ratio between the standard and the experimental arm and will be stratified by tumor stage and use of concurrent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to provide written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Biopsy proven diagnosis of squamous cell carcinoma of the oropharynx.
* Positive for HPV by p16 immunohistochemistry (IHC) or HPV in-situ hybridization (ISH)
* Clinical stage T1-3, N1 M0 (Stage I-II) as per AJCC 8th edition.
* Primary tumor < 30 cc
* Planned for curative chemoradiation
* For females of child-bearing age, a negative pregnancy test

Exclusion Criteria:

* Clinical N3 classification, as per AJCC 8th edition
* Clinically overt extranodal extension (ENE). As per AJCC 8th edition, clinically overt ENE is defined as invasion of the skin, infiltration of musculature/fixation to adjacent structures on clinical examination, cranial nerve, brachial plexus, sympathetic trunk or phrenic nerve invasion with dysfunction).
* Previous irradiation of the head and neck region
* Previous surgery of the HNC region (except for incisional or excisional biopsies)
* Pregnancy or breastfeeding
* Connective tissue disease
* Any medical condition that could, in the opinion of the investigator, prevent follow-up after radiotherapy.
* Non-Cisplatin concurrent chemotherapy
* Prior induction chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-02-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years after the end of chemoradiation
  Patient alive with no local, regional or distant recurrence at 2 years after the end of chemoradiation

SECONDARY OUTCOMES:
Subacute toxicity | Between 2 and 6 months after the end of chemoradiation
  Rate of grade ≥ 3 subacute toxicity
Acute toxicity | Less than 2 months after the end of chemoradiation
  Rate of grade ≥ 3 acute toxicity
Late toxicity | Between 6 months and 5-years after the end of chemoradiation
  Rate of grade ≥ 3 late toxicity
OS | At 2- and 5-years after the end of chemoradiation
  Overall survival
locoregional control | At 2- and 5-years after the end of chemoradiation
  Patient alive with locoregional control
Head and neck symptom burden | At baseline, and 1-, 3-, 6-, 12- months post-treatment, and yearly from years 2-5 after the end of chemoradiation
  Patient-reported head and neck symptom burden as measured by the MD Anderson Symptom Inventory Head and Neck Cancer Module. The core and head and neck cancer specific symptoms are rated on a 0-10 scale to indicate the presence and severity of the symptoms. Lower scores represent better functioning and quality of life.
Dysphagia | At baseline, and 1-, 3-, 6-, 12- months post-treatment, and yearly from years 2-5 after the end of chemoradiation
  Patient-reported dysphagia as measured by the MD Anderson Dysphagia Index. Overall score ranges from 0 to 100, with higher score representing better functioning and quality of life.
Time from treatment start to return to work | Measured in days and reported at 2-years post-treatment
  Time from first day of treatment start to first day of return to work.

CONTACTS AND LOCATIONS:
Overall Officials: Houda Bahig, MD PhD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Phuc-Felix Nguyen-Tan, MD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); David Palma, MD PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Jack Phan, MD PhD, Principal Investigator — M.D. Anderson Cancer Center; Khalil Sultanem, MD, Principal Investigator — Montreal Jewish General Hospital
Locations (2):
- Canada (2):
  - London Health Sciences Center, London, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No